CLINICAL TRIAL: NCT01654796
Title: Double-Blind, Proof-of-Concept (POC) Trial of Low Field Magnetic Stimulation (LFMS) Augmentation of Antidepressant Therapy in Treatment-Resistant Depression
Brief Title: Trial of Low Field Magnetic Stimulation Augmentation of Antidepressant Therapy in Treatment-Resistant Depression
Acronym: RAPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Yale University (Other); Icahn School of Medicine at Mount Sinai (Other); University of Texas Southwestern Medical Center (Other); University of Alabama at Birmingham (Other); Emory University (Other)
Responsible Party: Principal Investigator, Maurizio Fava, MD, Overall Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012P001233
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Treatment Resistant Depression
Keywords: Depression; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Field Magnetic Stimulation (Active Comparator): Patients in this arm will receive 2 days of active low field magnetic stimulation (LFMS) in phase 1, followed by 2 days of active low field magnetic stimulation (LFMS) in phase 2. LFMS is a novel, non-contact neuromodulation technique. LFMS is administered through a device while the patient lies on his/her back for 20 minutes.
  Interventions: Device: Low Field Magnetic Stimulation (LFMS)
- Sham (LFMS) (Placebo Comparator): Patients in this arm will receive 2 days of sham (not active) low field magnetic stimulation (LFMS) in phase 1, followed by 2 days of sham (not active) low field magnetic stimulation (LFMS) in phase 2.
  Interventions: Device: Sham LFMS
- Crossover Arm (Other): Patients in this group will receive two days of sham (not active) low field magnetic stimulation (LFMS) in phase 1, followed by two days of active low field magnetic stimulation (LFMS) in phase 2.
  Interventions: Device: Low Field Magnetic Stimulation (LFMS); Device: Sham LFMS

INTERVENTIONS:
Device: Low Field Magnetic Stimulation (LFMS) — The LFMS devices produces a unique magnetic field that may help alleviate symptoms of depression.
  Arms: Crossover Arm; Low Field Magnetic Stimulation
Device: Sham LFMS — Sham LFMS looks and sounds like the active treatment but does not produce any magnetic stimulation.
  Arms: Crossover Arm; Sham (LFMS)

SUMMARY:
This study is looking at the safety and efficacy of low field magnetic stimulation (LFMS) for treating patients with treatment resistant depression who are taking an antidepressant that is not working for them.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-65 years old
* Diagnosed with Major Depressive Disorder (MDD) and currently experiencing a Major Depressive Episode (MDE) of at least eight weeks
* A participant has Treatment Resistant Depression (TRD) of the current MDE
* Good general health
* For female participants, status of non-childbearing potential or use of an acceptable form of birth control
* Body mass index between 18-40 kg/m2
* Concurrent psychotherapy will be allowed if the type and frequency of the therapy has been stable for at least three months prior to screening and is expected to remain stable during participation in the study
* Concurrent hypnotic therapy will be allowed if the therapy has been stable for at least 4 weeks prior to screening and is expected to remain stable during the subject's participation in the study
* Participant must be able to lie flat for 20 minutes

Exclusion Criteria:

* A woman of childbearing potential who is not willing to use one of the specified forms of birth control during the study
* Pregnant or breastfeeding
* A woman with a positive pregnancy test at screening or baseline
* Participant has TRD of the current MDE with failure to achieve a satisfactory response, as perceived by the subject, to more than 3 treatment courses of a therapeutic dose of an antidepressant therapy of at least eight weeks duration
* Participant has a current diagnosis of a Substance Use Disorder with the exception of nicotine dependence, at screening or within six months prior to screening
* Current diagnosis of Axis I disorders other than Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Specific Phobia, Post Traumatic Stress Disorder or Complicated Grief (unless one of these is comorbid and clinically unstable, and/or the focus of the participant's treatment for the past six months or more).
* Subject has a history of schizophrenia or schizoaffective disorders, any history of psychotic symptoms or is on antipsychotic medication for the treatment of psychotic symptoms
* Subject has a history of eating disorders within five years of screening
* Subject has any Axis I or Axis II Disorder, which at screening is clinically predominant to their MDD or has been predominant at any time within six months prior to screening
* The participant is considered at significant risk for suicide during the study
* Subject has had electroconvulsive therapy in the current episode of depression
* Subject has had Transcranial Magnetic Stimulation or has received treatment with other experimental devices for the treatment of the current episode of depression
* Subject has received Vagus Nerve Stimulation at any time
* Dementia, delirium, amnestic, or other cognitive disorders
* There is a clinically significant abnormality on the screening physical examination
* Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation
* Known history or current episode of:

  --Uncontrolled hypertension, Recent myocardial infarction (within one year) or a history of more than one myocardial infarction, Syncopal event within the past year, Congestive heart failure, Angina pectoris
* Lifetime history of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system disorder (e.g., Alzheimer's or Parkinson's Disease), epilepsy, mental retardation, any other disease/procedure/accident/intervention associated with significant injury to or malfunction of the central nervous system, or a history of significant head trauma within the past two years.
* Lab abnormalities are present
* History of hypothyroidism and has been on a stable dosage of thyroid replacement medication for less than six months prior to screening
* Hisotry of hyperthyroidism which was treated (medically or sugically) less than six months prior to screening
* Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with the interpretation of study results
* History of positive screening urine test for drugs of abuse
* Patient with any non-removable stimulation device such as neurostimulators, pacemakers and cochlear implants
* Patients requiring treatment with excluded concomitant medications
* Patients who cannot be in a MRI
* Patients who are currently using a metal intrauterine device (IUD)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Iosifescu, MD, Principal Investigator — Mount Sinai School of Medecine; Gerald Sanacora, MD, Principal Investigator — Yale University; Madhukar Trivedi, MD, Principal Investigator — University of Texas; Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital (Coordinating Center); Mark Rapaport, MD, Principal Investigator — Emory University; Richard Shelton, MD, Principal Investigator — Univsity of Alabama at Birmingham; George I Papakostas, MD, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mount Sinai School of Medecine, New York, New York
  - University of Texas Southwestern, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Please note that while 85 subjects were randomized, only 84 subjects were included in the outcome analysis due to missing data. Adverse events are reported for all 85 subjects.
Groups:
- Sham LFMS First, Then Active LFMS: Patients in this group will receive two days of sham (not active) low field magnetic stimulation (LFMS) in phase 1, followed by two days of active low field magnetic stimulation (LFMS) in phase 2.
  Low Field Magnetic Stimulation (LFMS): The LFMS devices produces a unique magnetic field that may help alleviate symptoms of depression.
  Sham LFMS: Sham LFMS looks and sounds like the active treatment but does not produce any magnetic stimulation.
Period: Overall Study
Arm/Group | Low Field Magnetic Stimulation | Sham (LFMS) | Sham LFMS First, Then Active LFMS
Started | 26 | 29 | 29
Completed | 25 | 26 | 28
Not Completed | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Please note that while 85 subjects were randomized, only 84 subjects were included in the outcome analysis due to missing data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Field Magnetic Stimulation | Sham (LFMS) | Crossover Arm | Total
Number analyzed (Participants) | 26 | 29 | 29 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (14.8) | 50.7 (10) | 46.3 (14.6) | 48.3 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 15 | 47
  Male | 11 | 12 | 14 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 25 | 28 | 29 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 3 | 15
  White | 20 | 19 | 25 | 64
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression - 6 Items
Description: The total HAM-D-6 score is reported. The range of possible scores on the HAM-D-6 is from 0 to 22. Higher values indicate increased depression severity, and worse outcomes. This instrument is completed with a structured interview guide by the clinician based on his/her assessment of the patient's symptoms. This structured interview has been validated for use with time frames shorter than one week.The time frame for this scale is the past 24 hours.
Time Frame: Baseline and 48 hours after initiating treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Phase 1 Active LFMS: Participants in this group receive Active LFMS treatment for 2 days in Phase 1.
- Phase 1 Sham LFMS: Participants in this group received Sham LFMS treatment for 2 days in Phase 1.
- Phase 2 Active LFMS: Participants in this group received Active LFMS treatment for 2 days in Phase 2.
- Phase 2 Sham LFMS: Participants in this group received Sham LFMS treatment for 2 days in Phase 2.
Arm/Group | Phase 1 Active LFMS | Phase 1 Sham LFMS | Phase 2 Active LFMS | Phase 2 Sham LFMS
Number analyzed (Participants) | 26 | 58 | 18 | 21
units on a scale
  Baseline | 11.7 (2.2) | 11.3 (2.1) | 10.9 (2.2) | 9.4 (2.3)
  End of Phase | 8.8 (2.5) | 8.1 (3.7) | 9.6 (3.9) | 8.0 (3.7)
  Score Change | -2.8 (2.5) | -3.2 (3.3) | -1.3 (3.7) | -1.5 (2.4)

ADVERSE EVENTS:
Description: The adverse events listed include information for all 85 randomized subjects. Only 84 subjects were included in the outcome analysis due to missing data.
Arm/Group | Low Field Magnetic Stimulation | Sham (LFMS) | Crossover Arm
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 22/27 | 18/29 | 20/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Field Magnetic Stimulation (N=27) | Sham (LFMS) (N=29) | Crossover Arm (N=29)
Headache (Nervous system disorders) | 6 (9) | 10 (17) | 5 (7)
Dizziness (Vascular disorders) | 1 (2) | 2 (4) | 2 (2)
Irritability (Psychiatric disorders) | 2 (2) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 4 (4)
Blood Pressure Increased (Vascular disorders) | 0 (0) | 1 (4) | 1 (1)
Disturbance in Attention (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (3) | 2 (2)
Somnolence (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (2)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Hot Flush (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)
Memory Impairment (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Myalgia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Sleep Disorder (Psychiatric disorders) | 1 (2) | 1 (1) | 1 (1)
Abnormal Dreams (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Apathy (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Bruxism (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Electrocardiogram Abnormal (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Hiccups (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pain in Extremity (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Psychomotor Hyperactivity (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Toothache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain Lower (General disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drooling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Heart Rate Increased (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperlycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Libido Decreased (General disorders) | 1 (1) | 0 (0) | 0 (0)
Medial Tibial Stress Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myodesopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Obsessive-Compulsive Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Orgasm Abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0)
Parathyroid Tumor Benign (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus Congestion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Headache (General disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tension (General disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Weight Decreased (General disorders) | 1 (1) | 0 (0) | 0 (0)
Weight Increased (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No